CLINICAL TRIAL: NCT02779218
Title: Study of the Effects of the Combination of Motor Imagery Exercises and Transcranial Magnetic Stimulation (TMS) Type PAS in Patients After Hemiplegic Stroke
Brief Title: Combination of Motor Imagery Exercises and Brain Stimulation TMS Type PAS in Patients After Hemiplegic Stroke
Acronym: MIPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12 389 02
Record Dates: First submitted 2016-01-11; First posted 2016-05-20 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): The patients will receive in order :
  1. Paired Associative Stimulation
  2. Paired Associative Stimulation + Motor Imagery exercises
  3. Placebo Paired Associative Stimulation + Motor Imagery exercises
  Interventions: Procedure: Paired Associative Stimulation; Procedure: Paired Associative Stimulation + Motor Imagery exercises; Procedure: Placebo Paired Associative Stimulation + Motor Imagery exercises
- Sequence 2 (Experimental): The patients will receive in order :
  1. Paired Associative Stimulation + Motor Imagery exercises
  2. Placebo Paired Associative Stimulation + Motor Imagery exercises
  3. Paired Associative Stimulation
  Interventions: Procedure: Paired Associative Stimulation; Procedure: Paired Associative Stimulation + Motor Imagery exercises; Procedure: Placebo Paired Associative Stimulation + Motor Imagery exercises
- Sequence 3 (Experimental): The patients will receive in order :
  1. Placebo Paired Associative Stimulation + Motor Imagery exercises
  2. Paired Associative Stimulation
  3. Paired Associative Stimulation + Motor Imagery exercises
  Interventions: Procedure: Paired Associative Stimulation; Procedure: Paired Associative Stimulation + Motor Imagery exercises; Procedure: Placebo Paired Associative Stimulation + Motor Imagery exercises

INTERVENTIONS:
Procedure: Paired Associative Stimulation — Patient with Paired Associative Stimulation only
Procedure: Paired Associative Stimulation + Motor Imagery exercises — Patient with Paired Associative Stimulation + Motor Imagery exercises
Procedure: Placebo Paired Associative Stimulation + Motor Imagery exercises — Patient with placebo Paired Associative Stimulation + Motor Imagery exercises

SUMMARY:
Strokes represent, in industrialized countries the leading cause of acquired motor disability in adults older than 40. Stroke is responsible for France from 150 000 to 200 000 new cases of hemiplegia each year. These patients will see their deficit to improve during the first 6 months after stroke. This recovery is largely based on brain plasticity mechanisms and the rehabilitation has as main objective to optimize these mechanisms. However, only 20% of patients hospitalized in a rehabilitation sector recover a functional upper limb. This lack of functionality is not only due to overall strength gap but also to the predominance of this gap on the extension movements of the wrist and fingers.

Meanwhile, work on brain plasticity helped develop new techniques of non-invasive brain stimulation (Non-invasive Brain Stimulation, NIBS) as the model of coupled stimulations (Paired Associative Stimulation, PAS) for modulating way over effective brain plasticity. In previous studies, the investigators have shown over a 30 minutes session lasting facilitation (60mn) and specific motor evoked potential (MEP) of the Extensor Carpi Radialis (ECR). Several studies showed an adjuvant effect when GSIN were associated with learning of a motor task. For PAS, some studies have shown a greater facilitation when the latter is associated with muscle contraction.

The motor imagery (MI) is imagining a movement without realizing it, it is based on mechanisms similar to those of the real movement. This technique also showed its effects as an adjuvant therapy in hemiplegic patients, however, they remain lower than those obtained after a motor drive. Its use in patients with no motor makes its uniqueness and strength.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years
* Patients who have experienced a Stroke of more than one month
* Deficit out of the upper limb (Fugl Meyer member sup <50/66)
* Presence of ECR muscle MEP
* Able to carry the motor imagery according to a test by measuring chronometer
* Patient who signed informed consent
* Subject affiliated to the social security system

Exclusion Criteria:

* history of epilepsy or seizure
* MEP Lack of ECR
* Presence of a cons-indication for use of magnetic stimulation or MRI:

  * Surgical Clips, metal sutures, staples, stent
  * Osteosynthesis devices on the head or neck
  * Pacemaker
  * Implanted hearing aid
  * Ocular foreign body, shrapnel, bullets
  * Metal Worker
  * Heart Valve, endovascular equipment
  * Ventricular bypass valve
  * Pace-maker or neurostimulator
* Claustrophobia
* incapable adult Patient, safeguard justice, guardianship or trusteeship
* Pregnant women and / or breastfeeding (because lack of data in the literature regarding the absence of foetotoxic effect)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Effect of a reeducation session as assessed by amplitude of motor evoked potential | Day 1
  At the inclusion visit 25 minutes after stimulation
Effect of a reeducation session as assessed by amplitude of motor evoked potential | Week 1
  25 minutes after stimulation
Effect of a reeducation session as assessed by amplitude of motor evoked potential | Week 2
  25 minutes after stimulation
Effect of a reeducation session as assessed by amplitude of motor evoked potential | Week 3
  25 minutes after stimulation

SECONDARY OUTCOMES:
Resting Motor Threshold as assessed by minimal intensity to evoke a motor evoked potential | Week 1
  After the first stimulation
Resting Motor Threshold as assessed by minimal intensity to evoke a motor evoked potential | Week 2
  After the second stimulation
Resting Motor Threshold as assessed by minimal intensity to evoke a motor evoked potential | Week 3
  After the third stimulation
Active Motor Threshold as assessed by minimal intensity to evoke a motor evoked potential | Week 1
  After the first stimulation
Active Motor Threshold as assessed by minimal intensity to evoke a motor evoked potential | Week 2
  After the second stimulation
Active Motor Threshold as assessed by minimal intensity to evoke a motor evoked potential | Week 3
  After the third stimulation
Intensity curve as assessed by variation of intensity of motor evoked potential | Week 1
  After the first stimulation
Intensity curve as assessed by variation of intensity of motor evoked potential | Week 2
  After the second stimulation
Intensity curve as assessed by variation of intensity of motor evoked potential | Week 3
  After the third stimulation
Motricity of upper limb recovering as assessed by Fugl Meyer Score | Day 1
  After inclusion visit
Motricity of upper limb recovering as assessed by Fugl Meyer Score | Week 3
  After the third stimulation
Asymmetry index as assessed by resonance magnetic imaging | Day 1
  At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne CASTEL-LACANAL, MD, Principal Investigator — physical medecine and readaption
Locations (1):
- CHU Rangueil, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brihmat N, Tarri M, Gasq D, Marque P, Castel-Lacanal E, Loubinoux I. Cross-Modal Functional Connectivity of the Premotor Cortex Reflects Residual Motor Output After Stroke. Brain Connect. 2020 Jun;10(5):236-249. doi: 10.1089/brain.2020.0750. Epub 2020 Jun 11. PMID 32414294